CLINICAL TRIAL: NCT05131789
Title: Establishment and Application of Dementia Case Management Information System: A Preliminary Study - Phase 2
Brief Title: Establishment and Application of Dementia Case Management Information System: A Preliminary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Huei-Ling Huang, Associate Professor, PhD, RN, Department of Gerontology and Health Care Management, College of Nursing, Chang Gung University of Science and Technology, Taoyuan, Taiwan, R.O.C, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ZRRPF3L0041
Record Dates: First submitted 2021-10-31; First posted 2021-11-23 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Dementia
Keywords: Dementia; Case management; Information system
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Information System Group (Experimental): The dementia case managers in the experiment group use information system to perform case management.
  Interventions: Procedure: dementia case management information system

INTERVENTIONS:
Procedure: dementia case management information system — The investigators will develop an information system based on the data collected in our previous research, the content and method of dementia case management which will be established by the Delphi method, and then the dementia case management information system will be constructed accordingly.

SUMMARY:
The purpose of this study is to develop and examine the preliminary effects of an information system for facilitating dementia case management in the home setting.

This study is the second phase of the project. The first year is the development stage of the information system. In the second year, the investigators will conduct a pilot study to examine the effectiveness of the case management information system.

DETAILED DESCRIPTION:
The purpose of this study is to develop and examine the preliminary effects of an information system for facilitating dementia case management in the home setting. In the previous research (phase I), a mixed method was used to explore the content of case management and assess the needs of the information system.

This study is the second phase of the project. The first year is the development stage of the information system. Based on the data collected in the previous research (phase I), the content and method of dementia case management will be established by the Delphi method, and then the dementia case management information system will be constructed accordingly. In the second year, the investigators will conduct a pilot study to examine the effectiveness of the case management information system.

ELIGIBILITY:
Inclusion Criteria:

* Dementia Case Managers:

  1. Be at least 20 years old and could communicate in Chinese or Taiwanese.
  2. Currently work for dementia center, dementia care center, or Community-Based Dementia Care Center in Taiwan.
* Dementia family caregivers:

  1. Be at least 20 years old and could communicate in Chinese or Taiwanese.
  2. Primary caregivers
  3. The people with dementia under care are diagnosed with dementia Clinical Dementia Rating(CDR) 0.5 or higher.
  4. Live in northern Taiwan(including Taipei, New Taipei, Taoyuan, and Hsinchu).

Exclusion Criteria:

* Dementia Case Managers:

No longer working for dementia center, dementia care center, or Community-Based Dementia Care Center in Taiwan.

* Dementia family caregivers:

The people with dementia under care live in a long-term care facility or nursing home.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Dementia Care Professional Competency Assessment Scale | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Dementia Care Professional Competency at 1, 3, and 6 months.
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3). The scale is used to evaluate dementia care competency in dementia case managers (Huang et al., 2018).
  2. This Scale contains nine subscales (74 items), using Likert 5-point Likert scale from 1 to 5. A higher score means better competencies.
  3. This scale is used to evaluate the competence of dementia case managers.
Problem solving, Teamwork Competency Assessment Scale | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Problem solving, Teamwork Competency at 1, 3, and 6 months.
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3). There are 22 questions on this scale. The scale is used to evaluate the problem solving and teamwork competency of Dementia case managers. (Huang et al. 2018).
  2. This scale contains 22 items.10 items were used to evaluate problem solving competencies, 12 items were used to evaluate teamwork competencies. A higher score means better competencies.
  3. This scale is used to evaluate the competence of dementia case managers.
Caregiver Preparedness Scale - Professional version | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Caregiver Preparedness - Professional at 1,3, and 6 months.
  1. This scale was developed by our research team by referring to The Preparedness for Caregiving Scale (PCS) developed by Archbold et al. This scale is to rate how well prepared they believe they are for caregiving (Archbold et al.,1990; Huang, Kuo, et al., 2013).
  2. This 11-items scale was scored on a 5-point Likert scale from 1 (unprepared) to 5 (well prepared). Scores range from 11 to 55, with higher scores representing greater preparedness for caregiving tasks. A final question is an open-end question.
  3. This scale is used to evaluate the competence of dementia case managers.
Basic information of dementia and family caregivers | The investigators will evaluate before the intervention.
  1. The persons with dementia include age, gender, education level, marital status, degree of dementia, period of illness, Mini-Mental State Examination (MMSE), etc. The family caregivers include age, gender, education level, marital status, etc.
  2. This scale is used to evaluate family caregivers.
Cohen-Mansfield Agitation Inventory (CMAI) | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline behavioral problems (CMAI) at 1, 3, and 6 months.
  1. Dementia's behavioral problems were measured by the Chinese version of the CMAI, community form (Cohen-Mansfield, J et al. 1989, 1991, C.K.Y. Lai, pers. comm.).
  2. The 43-item CMAI has four subscales that assess four groups of behavioral problems: physically non-aggressive behavior, physically aggressive behavior, verbally aggressive behavior and verbally non-aggressive behavior. Each item's score ranges from 1 (never happened) to 7 (several times in an hour). Scores can range from 43-301, with higher scores representing more frequent or more types of behavioral problems.
  3. This scale is used to evaluate family caregivers.
Agitation Management Self-Efficacy Scale (AMSS) | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline caregiver self-efficacy to handle behavioral problems (AMSS) at 1, 3, and 6 months.
  1. Family caregivers' self-efficacy for caring agitated behavior of older people with dementia was measured by the Agitation Management Self-Efficacy Scale (AMSS), which was developed by our research team. (Huang, Shyu, Chen, & Hsu, 2009)
  2. For each of the 43 behavioral problems identified by the Chinese version of the CMAI, caregivers are asked how confident they feel about handling the problem. Each AMSS item is scored on a Likert-type scale from 1 (not able to handle at all) to 5 (totally able to handle). Total scores range from 43-215. Higher scores represent greater caregiver self-efficacy to handle behavioral problems.
  3. This scale is used to evaluate family caregivers.
Activities of daily living (ADL) | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline ADL at 1, 3, and 6 months.
  1. García-Casal JA, Loizeau A, Csipke E, Franco-Martín M, Perea-Bartolomé MV, Orrell M. Computer-based cognitive interventions for people living with dementia: a systematic literature review and meta-analysis. Aging Ment Health.2016; 25: 1-14.
  2. The ADL refers to activities oriented toward taking care of one's own body.
  3. This scale assesses 10 items related to the activity including feeding, transfer, grooming, toilet use, bathing, mobility, stairs, dressing, bowels, and bladder. Each item is scored from 0 (maximum disability and dependency) to 20 (maximum strength and independence). Scores can range from 0 to 100, with higher scores representing more independence.
  4. This scale is used to evaluate family caregivers.
Instrumental Activities of Daily Living (IADL) | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline IADL at 1, 3, and 6 months.
  1. Ryu SY, Lee SB, Kim TW, Lee TJ. Subjective memory complaints, depressive symptoms and instrumental activities of daily living in mild cognitive impairment. Int Psychogeriatr. 2015; 11: 1-8.
  2. The IADL refers to activities oriented toward interacting with the environment and that are often complex-generally optional in nature.
  3. This scale assesses 8 items related to the activity including the ability to use a phone, shopping, the model of transportation, meal preparation, housekeeping, laundry, the responsibility for owns medication, and the ability to handle finance. Each item is scored from 0 (dependency) to 3 (independence). Scores can range from 0 to 24, with higher scores representing more independence.
  4. This scale is used to evaluate family caregivers.
Caregiver competence Scale | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Caregiver competence at 1, 3, and 6 months.
  1. This scale was developed by our research team by referring to The measure of caregiver competence developed by Kosberg and Cairl. (Kosberg & Cairl, 1991; Huang & Shyu, 2003)
  2. This scale is used to assess the caregiver's ability to perform care tasks.
  3. Each item is scored from 1 to 5. Scores can range from 20 to 100, with higher scores representing the ability better.
  4. This scale is used to evaluate family caregivers.
Caregiver Preparedness Scale - family caregiver version | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Caregiver Preparedness - family caregiver at 1, 3, and 6 months.
  1. This scale was developed by our research team by referring to The Preparedness for Caregiving Scale (PCS) developed by Archbold et al. This scale is to rate how well prepared they believe they are for caregiving (Archbold et al.,1990; Huang, Kuo, et al., 2013).
  2. This 11-items scale was scored on a 5-point Likert scale from 1 (unprepared) to 5 (well prepared). Scores range from 11 to 55, with higher scores representing greater preparedness for caregiving tasks. A final question is an open-end question.
  3. This scale is used to evaluate family caregivers.
36-item short-form health survey (SF-36) | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline quality of life (SF-36) at 1, 3, and 6 months.
  1. Ware J. E., & Sherbourne, C. D. (1992). The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Medical care, 473-483.
  2. The SF-36 measures eight scales, with higher scores representing the greater quality of life.
  3. This scale is used to evaluate family caregivers.
Qualitative interview | The investigators will conduct qualitative interviews before the intervention, and after intervention for 1 month.
  Conduct qualitative interviews with dementia case managers, focusing on the use of information system.

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Ling Huang, PhD, Study Chair — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan